CLINICAL TRIAL: NCT05694065
Title: Functional ComprEhensive AssessmenT by Intravascular UltrasoUnd Reconstruction in Patients With Suspected IschEmic Coronary Artery Disease (FEATURE)
Brief Title: Functional ComprEhensive AssessmenT by IVUS Reconstruction in Patients With Suspected IschEmic Heart Disease (FEATURE)
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: School of Biomedical Engineering, Shanghai Jiao Tong University (Unknown); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20221110025331724
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigating the diagnostic accuracy of online Ultrasonic Flow Ratio (UFR) assessment to identify hemodynamically significant coronary stenosis in patients with suspected ischemic heart disease using angiography-derived fractional flow reserve (FFR) as a reference standard.

DETAILED DESCRIPTION:
1. Study overview This is a prospective, single-center, observational registry study of patients with suspected ischemic coronary artery disease. The purpose of this registry is to investigate the accuracy of online UFR assessment to identify hemodynamically significant coronary stenosis in patients with suspected ischemic heart disease using angiography-derived FFR as a reference standard.
2. Study population and sample size calculation are based on the diagnostic performance of previous studies, where an accuracy of 92% was found for UFR. Investigators conservatively estimate the diagnostic accuracy of online UFR assessment as 90% for consecutively enrolled patient population, and with a test target value set as 78% at a two-side significance level of 0.05, statistical power as 90%. Considering incomplete FFR/UFR data of 10% at most, a total of 112 patients need to be enrolled.
3. Participant enrollment was completed in November 2024; the study is currently in the follow-up phase with ongoing data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years
* Patients suspected with ischemic heart disease
* ≥ 1 diseased vessel with angiographic percent diameter stenosis between 40% and 80% in a vessel ≥ 2.5mm by visual estimation
* Target vessels are limited to major epicardial coronary arteries (left anterior descending artery [LAD], left circumflex artery [LCX], right coronary artery [RCA])

Exclusion Criteria:

* Patients with previous coronary artery bypass grafting (CABG)
* Myocardial infarction within 72h of coronary angiography
* Allergy to the contrast agent or adenosine
* Left main coronary artery stenosis ≥ 50%
* Target vessel with in-stent restenosis
* Target vessel with severe tortuosity or angulation
* 100% occlusion of target vessel
* Target vessel spasm or injury
* Target vessel with severe myocardial bridge
* Target vessel with severe thrombosis
* Intravascular ultrasound (IVUS) pullback fails to cover the complete target lesion
* Presence of false lumen at target vessel based on IVUS
* A serum creatinine level >150 umol/l, or a glomerular filtration rate < 45 ml/kg/1.73 m^2
* Heart failure
* Ineligible for diagnostic intervention (IVUS or FFR examination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected ischemic heart disease who undergo coronary angiography.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Ding, MD, PhD, Principal Investigator — Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Assessment in Patients With Suspected Ischemic Heart Disease: Onsite Ultrasonic Flow Ratio (UFR) and Fractional Flow Reserve (FFR) Assessment in Patients with Suspected Ischemic Heart Disease
Period: Overall Study
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Started | 112
Completed | 106
Not Completed | 6
Not completed — Intravascular ultrasound (IVUS) pullback fails to cover the complete target lesion | 3
Not completed — Ineligible for diagnostic intervention (IVUS or FFR examination) | 2
Not completed — Target vessel with severe myocardial bridge | 1

BASELINE CHARACTERISTICS:
Groups:
- Functional Assessment in Patients With Suspected Ischemic Heart Disease: Onsite UFR and FFR Assessment in Patients with Suspected Ischemic Heart Disease
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Six participants were excluded according to the predefined exclusion criteria.
  years | 68.5 [57.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Six participants were excluded according to the predefined exclusion criteria.
  Participants
    Female | 30
    Male | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Population: Six participants were excluded according to the predefined exclusion criteria.
  Kg/m^2 | 24.6 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of Onsite UFR
Description: UFR was computed as the pressure ratio across a coronary stenosis, using FFR ≤0.80 as the reference standard for hemodynamically significant stenosis.
  The diagnostic performance of onsite UFR was assessed by the area under the receiver operating characteristic (ROC) curve analysis, with diagnostic accuracy defined as the percentage of all correctly classified cases (true positives and true negatives) in the total population.
Time Frame: baseline
Population: Six participants were excluded according to the predefined exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of correctly classified cases
Groups:
- Functional Assessment in Patients With Suspected Ischemic Heart Disease: FFR and UFR were assessed onsite in the catheterization laboratory for patients with suspected ischemic heart disease.
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
percentage of correctly classified cases | 94 [88 to 97]
Statistical Analysis 1: Comparison: Functional Assessment in Patients With Suspected Ischemic Heart Disease; Test type: Other; The diagnostic discrimination ability of UFR was analyzed by ROC curve analysis using the DeLong method. Cutoff value of ≤0.80 was used for FFR and UFR to define the physiological significance of a coronary stenosis, with two-sided P<0.05 considered statistically significant

2. Secondary Outcome: Sensitivity of Onsite UFR
Description: The diagnostic performance of onsite UFR was assessed by ROC curve analysis, using an FFR ≤0.80 as the reference standard.
  Sensitivity was defined as the percentage of true positives correctly identified by UFR.
Time Frame: baseline
Population: Six participants were excluded according to the predefined exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
percentage of true positives | 88 [75 to 96]

3. Secondary Outcome: Specificity of Onsite UFR
Description: The diagnostic performance of onsite UFR was assessed by ROC curve analysis, using an FFR ≤0.80 as the reference standard.
  Specificity was defined as the percentage of true negatives correctly identified by UFR.
Time Frame: baseline
Population: Six participants were excluded according to the predefined exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
percentage of true negatives | 97 [90 to 99]

4. Secondary Outcome: Sensitivity of Minimal Lumen Area (MLA)
Description: The diagnostic performance of MLA was assessed by ROC curve analysis, using an FFR ≤0.80 as the reference standard.
  Sensitivity was defined as the percentage of true positives correctly identified by the prespecified MLA cutoff value.
Time Frame: baseline
Population: Six participants were excluded according to the predefined exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
percentage of true positives | 47 [31 to 62]

5. Secondary Outcome: Specificity of MLA
Description: The diagnostic performance of MLA was assessed by ROC curve analysis, using an FFR ≤0.80 as the reference standard.
  Specificity was defined as the percentage of true negatives correctly identified by the prespecified MLA cutoff value.
Time Frame: baseline
Population: Six participants were excluded according to the predefined exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
Number analyzed (Participants) | 106
percentage of true negatives | 84 [75 to 91]
Statistical Analysis 1: Comparison: Functional Assessment in Patients With Suspected Ischemic Heart Disease; Test type: Other; The diagnostic discrimination abilities of UFR and MLA were compared by ROC curves analysis using the DeLong method. A prespecified MLA cutoff value was applied based on the prior study. Cutoff value of ≤0.80 was used for FFR and UFR to define the physiological significance of a coronary stenosis, with two-sided P<0.05 considered statistically significant

ADVERSE EVENTS:
Time Frame: Not monitored as this is a prospective observational study without any intervention.
Description: Adverse events were not systematically collected or assessed as primary or secondary outcomes in this observational study protocol.
Arm/Group | Functional Assessment in Patients With Suspected Ischemic Heart Disease
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT05694065/Prot_SAP_000.pdf